CLINICAL TRIAL: NCT03537027
Title: Comparing the Efficiency of Vitamin D3 and 25-hydroxyvitamin D3 Treatment on Changes of the Transcriptome of Low Vitamin D Responders
Brief Title: Efficiency of Vitamin D3 and 25-hydroxyvitamin D3 on Transcriptomic Changes of Low Vitamin D Responders
Acronym: VitDHiD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Carsten Carlberg, Professor of biochemistry, University of Eastern Finland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VitDHiD
Record Dates: First submitted 2018-04-26; First posted 2018-05-25 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Vitamin D Receptor Target Gene Expression; Serum 25(OH)D Concentration
Keywords: vitamin D3; cholecalciferol; calcidiol; 25-hydroxyvitamin D; gene expression; vitamin D receptor; adults; clinical trial
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D3 (Experimental): 2000 micrograms of vitamin D3 in two doses during one day
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — In total 20 pills will be taken by the subjects, each containing 100 micrograms of vitamin D3, resulting in the total amount of 2000 micrograms of vitamin D3. Of the 20 pills, 10 will be taken in the morning with breakfast and 10 with lunch.
  Other Names: cholecalciferol

SUMMARY:
The purpose of the study is to investigate in vivo whether a high-dose vitamin D3 oral bolus (2000 micrograms) produces marked vitamin D receptor target gene expression response and whether there is large inter-individual variation. These effects are compared to in vitro treatment of peripheral blood mononuclear cells from these subjects with 25(OH)D.

DETAILED DESCRIPTION:
Serum 25-hydroxyvitamin D3 [25(OH)D3] is a well-established marker for vitamin D status of the human body. In addition to the general importance of vitamin D for bone health, low serum 25(OH)D3 concentrations have been associated with increased risk of several health outcomes, such as autoimmune diseases, type 2 diabetes and cardiovascular complications. However, there is significant inter-individual variation in the average serum 25(OH)D3 concentrations and also in the response to supplementation with vitamin D. Genetic and epigenetic factors have been suggested to be responsible for a large part of the variation, but currently there is little information about the health effects of the variation.

In our previous studies VitDmet (Clinicaltrials.gov NCT01479933) and VitDbol (Clinicaltrials.gov NCT02063334) we showed that the participants can be classified into high, mid and low responders to vitamin D and defined the new biomarker "vitamin D response index". Some 25% of the population seem to be low responders and are under higher risk to suffer from insufficient supplementation with vitamin D. The current study will focus on low vitamin D responders (among the 40 healthy individuals recruited in the study, 20-60 years old), i.e. it will use the same oral vitamin D3 bolus (2,000 µg, i.e. 80,000 IU in one day) as in our VitDbol study, in order to identify low vitamin D responders.

By in vitro treatment of peripheral blood mononuclear cells (PBMCs) of low responders with 25(OH)D3 for 24 h (in comparison to in vitro stimulations with 1,25-dihydroxyvitamin D3 [1,25(OH)2D3] and in vivo vitamin D3 supplementation of the same subjects) we will obtain samples that allow the transcriptome-wide investigation of changes in gene expression. The underlying hypothesis of this study is that a stimulation with 25(OH)D3 is more efficient than a treatment with vitamin D3, so that in future low vitamin D responders may be supplemented with 25(OH)D3 rather than with vitamin D3.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* BMI 20-25 kg/m2.

Exclusion Criteria:

* History of kidney stones, renal failure or dialysis, hypercalcemia, hypo- or hyperparathyroidism, severe liver disease (cirrhosis), or sarcoidosis or other granulomatous diseases, such as active chronic tuberculosis or Wegener's granulomatosis.
* Continuous use of anti-inflammatory medicines.
* Regular use of supplements containing over 20 micrograms of vitamin D.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
In vivo change from baseline in vitamin D target gene expression in the subjects | 24 hours after the baseline
  Effect of 2000 microgram vitamin D3 dose on the expression of vitamin D receptor target genes
In vitro change from baseline in vitamin D target gene expression in peripheral blood mononuclear cells | 24 hours after the baseline
  Effects of treatment of cells for 24 h with 100 nM of 25(OH)D3, 1 nM of 1,25(OH)2D3 or vehicle (solvent) on the expression of vitamin D receptor target genes

SECONDARY OUTCOMES:
In vivo change from baseline in serum 25(OH)D concentration | 24 hours after the baseline
  Effect of 2000 microgram vitamin D3 dose on serum 25(OH)D3 concentrations
In vivo change from baseline in serum calcium concentration (safety and tolerability) | 24 hours after the baseline
  Effect of 2000 microgram vitamin D3 dose on in vivo changes in serum calcium concentrations
In vivo change from baseline in serum alanine transaminase concentration (safety and tolerability) | 24 hours after the baseline
  Effect of 2000 microgram vitamin D3 dose on in vivo changes in serum alanine transaminase (ALAT) concentrations
In vivo change from baseline in serum gamma-glutamyl transferase concentration (safety and tolerability) | 24 hours after the baseline
  Effect of 2000 microgram vitamin D3 dose on in vivo changes in serum gamma-glutamyl transferase (GGT) concentrations
In vivo change from baseline in serum creatinine concentration (safety and tolerability) | 24 hours after the baseline
  Effect of 2000 microgram vitamin D3 dose on in vivo changes in serum creatinine concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Carlberg, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No